CLINICAL TRIAL: NCT02976194
Title: Intraocular Cytokine Changes in Recurrence of Polypoidal Choroidal Vasculopathy
Brief Title: Intraocular Cytokine in Recurrence of Polypoidal Choroidal Vasculopathy
Acronym: CyPov
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pusan National University Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-0186
Record Dates: First submitted 2016-11-22; First posted 2016-11-29 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Exudative Age-related Macular Degeneration; Polypoidal Choroidal Vasculopathy
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pro-re-nata (Experimental): Ranibizumab 0.5mg is injected in to the vitreous cavity. An injection is given every 4 weeks three times, and then the patient will be followed up every 4 weeks. An addition injection is given as needed. Recurrence is defined as increase of exudative changes, or increase of 10% or more in central subfield macular thickness (CSMT) measured using optical coherence tomography. Aqueous humor is sampled from the anterior chamber before injection at baseline, 8 weeks and 20 weeks.
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — Ranibizumab 0.5mg is injected into the vitreous cavity through the pars plana using 30 gauge (or narrower) needle-attached syringe.
  Other Names: Lucentis

SUMMARY:
Changes of intraocular cytokines including vascular endothelial growth factor (VEGF) will be measured in recurrence of polypoidal choroidal vasculopathy (PCV) during treatment of ranibizumab.

DETAILED DESCRIPTION:
PCV is regarded as a subtype of age-related macular degeneration (ARMD), but has several different features such as polypoidal terminal of new vessels, and relative resistance to anti-VEGF treatment. Other cytokines then VEGF are thought to be associated with development and progression of the disease. The aim of the this study is to investigate intraocular cytokines related to recurrence of polypoidal choroidal vasculopathy. Aqueous humor will be sampled from the anterior chamber at baseline, after loading injections of ranibizumab and at recurrence. The concentration of various cytokines will be measured in the aqueous humor.

ELIGIBILITY:
Inclusion Criteria:

1. Submacular PCV diagnosed based on branching neovascular networks having polypoidal dilatation in ICGA.
2. Presence of exudative changes involving the fovea in OCT
3. Decreased visual acuity to 20/320 - 20/40 to be primarily the results of PCV in the study eye.
4. Willing and able to comply with clinic visits and study-related procedures, and provide a signed informed consent form.

Exclusion Criteria:

1. Extramacular PCV.
2. Presence of pathologic changes blocking 50% or more area of the lesion in angiography.
3. Any anti-VEGF treatment in the study eye within 180 days of day 1.
4. Previous photodynamic therapy in the study eye.
5. History of intraocular surgery except uncomplicated cataract surgery performed before 90 days or more from day 1.
6. Presence of exudative ARMD requiring anti-VEGF treatment in the other eye.
7. Presence of other ocular disease that may compromise visual acuity in the study eye.
8. Uncontrolled systemic disease.
9. Active intraocular or periocular infection.
10. Active intraocular inflammation.
11. Hypersensitivity to ranibizumab or excipients.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2016-11-22 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Changes of VEGF-A from 8 weeks to 20 weeks | 8 weeks and 20 weeks
  Intraocular concentration of VEGF-A is measured using multiplex immunoassay.

SECONDARY OUTCOMES:
Changes of the other cytokines from 8 weeks to 20 weeks | 8 weeks and 20 weeks
  Intraocular concentration of the other cytokines including angiopoietin-1, interleukin-10 (IL-10), platelet-derived growth factor (PDGF) and placental growth factor (PlGF) is measured using multiplex immunoassay.
Changes of cytokines from baseline to 8 weeks | baseline and 8 weeks
  Intraocular concentration of cytokines including VEGF, angiopoietin-1, IL-10, PDGF and PlGF is measured using multiplex immunoassay.
Correlation between time to recurrence and cytokine concentration at baseline and 8 weeks. | baseline and 8 weeks
  Time to recurrence is defined as number of weeks from 8 to recurrence. The correlation is assessed using non-parametric analysis, or Spearman's ranked correlation.
Correlation between vision changes and cytokine concentration changes | baseline and 24 weeks.
  Visual acuity is assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart. The ETDRS chart includes 100 letters as the maximum possible score, and 0 letters read as the minimum possible score. Visual acuity of 85 letters is equivalent to 20/20. Higher score represents better functioning. The correlation is assessed using non-parametric analysis, or Spearman's ranked correlation.
Correlation between CSMT and cytokine concentration | baseline, 8 weeks and 20 weeks.
  CSMT is central 1mm thickness of the macula measured using spectral-domain optical coherence tomography (OCT). Normal thickness is around 250μm. Increased CSMT is regarded as increase of en exudative sign. The correlation is assessed using non-parametric analysis, or Spearman's ranked correlation.
Correlation between choroidal thickness and cytokine concentration | baseline, 8 weeks and 20 weeks.
  Choroidal thickness is thickness of the choroid measured at the foveal center using spectral-domain OCT. Increased choroidal thickness was reported to be related to poor response to anti-VEGF treatment. The correlation is assessed using non-parametric analysis, or Spearman's ranked correlation.
Correlation between area of new vessels and cytokine concentration | baseline
  Area of new vessels is measured in indocyanine green angiography (ICGA) obtained at baseline. The correlation is assessed using non-parametric analysis, or Spearman's ranked correlation.
Correlation between polyp closure and cytokine concentration changes | baseline and 8 weeks
  Polyp closure is defined as disappearance of polypoidal terminal in new vessels assessed in ICGA at 8 weeks. The difference of cytokine concentration is assessed between the closed group and un-closed group using non-parametric analysis, or Mann-Whitney U test.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Eun Lee, MD, PhD, Principal Investigator — Pusan National University Hospital
Locations (2):
- South Korea (2):
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Pusan National University Hospital, Busan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cha DM, Woo SJ, Kim HJ, Lee C, Park KH. Comparative analysis of aqueous humor cytokine levels between patients with exudative age-related macular degeneration and normal controls. Invest Ophthalmol Vis Sci. 2013 Oct 25;54(10):7038-44. doi: 10.1167/iovs.13-12730. PMID 24106111
- [Background] Rezar-Dreindl S, Sacu S, Eibenberger K, Pollreisz A, Buhl W, Georgopoulos M, Krall C, Weigert G, Schmidt-Erfurth U. The Intraocular Cytokine Profile and Therapeutic Response in Persistent Neovascular Age-Related Macular Degeneration. Invest Ophthalmol Vis Sci. 2016 Aug 1;57(10):4144-50. doi: 10.1167/iovs.16-19772. PMID 27537264
- [Background] Hu J, Leng X, Hu Y, Atik A, Song X, Li Z, Liu Y, Lu L. The Features of Inflammation Factors Concentrations in Aqueous Humor of Polypoidal Choroidal Vasculopathy. PLoS One. 2016 Jan 22;11(1):e0147346. doi: 10.1371/journal.pone.0147346. eCollection 2016. PMID 26799405
- [Background] Sakurada Y, Nakamura Y, Yoneyama S, Mabuchi F, Gotoh T, Tateno Y, Sugiyama A, Kubota T, Iijima H. Aqueous humor cytokine levels in patients with polypoidal choroidal vasculopathy and neovascular age-related macular degeneration. Ophthalmic Res. 2015;53(1):2-7. doi: 10.1159/000365487. Epub 2014 Nov 29. PMID 25472810
- [Background] Tong JP, Chan WM, Liu DT, Lai TY, Choy KW, Pang CP, Lam DS. Aqueous humor levels of vascular endothelial growth factor and pigment epithelium-derived factor in polypoidal choroidal vasculopathy and choroidal neovascularization. Am J Ophthalmol. 2006 Mar;141(3):456-62. doi: 10.1016/j.ajo.2005.10.012. PMID 16490490